CLINICAL TRIAL: NCT02115256
Title: Intravenous Terbutaline Versus Intravenous Nitroglycerine for External Cephalic Version: A Double-Blinded Randomized Controlled Trial in Nulliparous Women
Brief Title: Study to Evaluate is ECV Success is Improved and the Side Effects Reduced With the Use of IV NTGL Versus Terbutaline
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficult recruitment
Sponsor: Yaakov Beilin (Other)
Responsible Party: Sponsor-Investigator, Yaakov Beilin, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-0636
Record Dates: First submitted 2014-04-13; First posted 2014-04-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: External Cephalic Version
Keywords: External Cephalic Version; breech
MeSH Terms: interventions — Terbutaline; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Terbutaline (Active Comparator): 0.25 mL of Intravenous Terbutaline
  Interventions: Drug: Intravenous Terbutaline
- Intravenous Nitroglycerine (Active Comparator): IV nitroglycerine 100 micrograms three minutes before beginning the procedure, then followed by a second dose 3 minutes later just after the start of the procedure for a total of 200 micrograms.
  Interventions: Drug: Intravenous Nitroglycerine

INTERVENTIONS:
Drug: Intravenous Terbutaline — 0.25 mL of Intravenous Terbutaline. This will be followed 3 minutes later by an injection of 0.25 mL IV of normal saline.
  Other Names: Terbutaline; Brethine; Bricanyl; Brethaire; Terbutalin; (RS)-5-[2-(tert-butylamino)-1-hydroxyethyl]benzene-1,3-diol)
  Arms: Intravenous Terbutaline
Drug: Intravenous Nitroglycerine — The dose of IV nitroglycerine will be 100 micrograms three minutes before beginning the procedure, and because of it's short half-life (approximately 3 minutes) will be followed by a second dose 3 minutes later just after the start of the procedure for a total of 200 micrograms.
  Other Names: Nitroglycerine; Nitroglycerin; Trinitroglycerin; Trinitroglycerine; nitro; 1,2,3-trinitroxypropane
  Arms: Intravenous Nitroglycerine

SUMMARY:
Breech presentation of a term pregnancy is a common occurrence. A procedure known as external cephalic version (ECV) is frequently used by obstetricians to turn the baby into the vertex position prior to delivery in order to avoid a cesarean section and the associated risks. Medications to relax the uterus, known as tocolytics, are used in conjunction with the procedure as they have been shown to improve the success rate of ECV, but with inconsistent, varying results.

DETAILED DESCRIPTION:
Breech presentation occurs in approximately 3-4% of all births and all women with breech presentation at term undergo cesarean delivery. The only way to avoid a cesarean is to manually turn the baby prior to the date of delivery, a procedure known as elective external cephalic version (ECV). ECV has been shown to reduce the frequency of breech presentation at term and thus lessen the risks associated with breech delivery and those of cesarean section, with little risk to the mother or baby. Tocolysis, administered immediately prior to the ECV and commonly used at The Mount Sinai Hospital, has been shown to improve the success rate of ECV. Several different agents are known to cause tocolysis. These include beta-mimetics (ritodrine, terbutaline), nitroglycerine (NTGL) and nifedipine.Terbutaline has been shown to improve success rate of ECV. Another study published in 2004 by El-Sayed et al showed that subcutaneous terbutaline was associated with higher rates of successful ECV than IV NTGL in term patients. There is inconsistent data in regard to the success rate of ECV with NTGL. In a study published in 2003 by Bujold et al, NTGL was associated with a higher rate of side effects and a lower rate of successful ECV when compared to ritodrine. Another study published in 2009 by Hilton et al showed that NTGL was more efficacious for ECV in nulliparous versus multiparous women. Yet another study published in 2009 by Yanny et al showed no differences between sublingual NTGL versus placebo in efficacy, and reported no significant side effects. A study published in 2003 by Bujold et al showed that sublingual NTGL was associated with a higher incidence of headache and did not improve the success rate of ECV. It may be beneficial to use NTGL instead of terbutaline because NTGL is a shorter acting agent and the procedure itself only lasts 10-15 minutes. Additionally, both medications have side effects. Terbutaline is associated with maternal tachycardia, hyperglycemia, hypokalemia, pulmonary edema, cardiac arrhythmias, hypertension and myocardial ischemia, and NTGL is associated with maternal nausea, vomiting, headache, and hypotension. For both medications the side effects are self- limiting but depending on the patient's co-morbidities one drug may be beneficial for that individual patient.

To date no study has compared the efficacy of intravenous terbutaline versus intravenous NTGL in women presenting for ECV. The purpose of this study is to determine if the success rate of ECV can be improved with the use of IV NTGL.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18-35 years of age
* 37 weeks gestation
* Breech presentation

Exclusion Criteria:

* Patients with ruptured membranes
* Multiple gestation
* Maternal age (age > 35)
* With known medical comorbidities (including hypertension (HTN), arrhythmias, endocrinologic diseases such as diabetes and thyroid disease, scoliosis, asthma)
* Allergies to nitroglycerine or terbutaline
* Prior abdominal or uterine surgery

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Beilin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 Participants were enrolled from 06/12/2014 to 05/12/2015.
Period: Overall Study
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (1) | 36 (2) | 34 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Successful Version of the Fetus Into the Vertex Position
Description: Number of participants that had successful version of the fetus into the vertex position.
Time Frame: average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
Number analyzed (Participants) | 3 | 2
Participants | 3 | 0

2. Secondary Outcome: Hypotension
Description: Number of participants with hypotension
Time Frame: average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
Number analyzed (Participants) | 3 | 2
Participants | 2 | 1

3. Secondary Outcome: Need for Cesarean Delivery
Description: Number of participants that needed a cesarean delivery
Time Frame: average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

4. Secondary Outcome: Tachycardia
Description: Number of participants that had tachycardia
Time Frame: average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
Number analyzed (Participants) | 3 | 2
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Terbutaline | Intravenous Nitroglycerine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes